CLINICAL TRIAL: NCT04247347
Title: Tailored Health Self-Management Interventions for Highly Distressed Caregivers: Family Members of Persons With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Jaclene A. Zauszniewski, Principal Investigator, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3R01NR01S817-04S1
Record Dates: First submitted 2020-01-24; First posted 2020-01-30 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Stress; Carer Stress Syndrome; Dementia; Alzheimer Disease
Keywords: Caregiver; Biofeedback; Resourcefulness; Self-Management
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Resourcefulness Training (Experimental): A cognitive-behavioral intervention presented within an audiovisual format using a tablet computer that consists of teaching and reinforcing personal (self-help) and social (help-seeking) resourcefulness skills.
  Interventions: Behavioral: Resourcefulness Training
- Dementia Education (Active Comparator): An educational program designed to teach family caregivers about the characteristics, types, causes, and risk factors of dementia, as well as teach about health promotion, the stages of dementia, behavior changes, communicating with a family member with dementia, and caring for oneself. The content to be presented within an audiovisual format using a tablet computer follows recommendations and guidelines developed through research and by the Alzheimer's Association and the National Institute on Aging.
  Interventions: Other: Dementia Education
- Biofeedback Training (Experimental): Use of a heart-rate variability (HRV) tracking device to enable one to learn to alter physiology to improve health. Devices are used to measure physiological activity, e.g., breathing and heart function, and provide rapid, accurate "feedback" to the user, thereby enabling desired physiological changes that can endure over time without continued use of the device and to continue to influence behavior.
  Interventions: Behavioral: Biofeedback Training

INTERVENTIONS:
Behavioral: Biofeedback Training — Use of a heart-rate variability (HRV) tracking device to enable one to learn to alter physiology to improve health. Devices are used to measure physiological activity, e.g., breathing and heart function, and provide rapid, accurate "feedback" to the user, thereby enabling desired physiological changes that can endure over time without continued use of the device and to continue to influence behavior.
  Arms: Biofeedback Training
Other: Dementia Education — An educational program designed to teach family caregivers about the characteristics, types, causes, and risk factors of dementia, as well as teach about health promotion, the stages of dementia, behavior changes, communicating with a family member with dementia, and caring for oneself. The content to be presented within an audiovisual format using a tablet computer follows recommendations and guidelines developed through research and by the Alzheimer's Association and the National Institute on Aging.
  Arms: Dementia Education
Behavioral: Resourcefulness Training — A cognitive-behavioral intervention presented within an audiovisual format using a tablet computer that consists of teaching and reinforcing personal (self-help) and social (help-seeking) resourcefulness skills.
  Arms: Resourcefulness Training

SUMMARY:
How do different health self-management interventions (resourcefulness training or biofeedback training) compare to usual care (dementia education) in affecting the health risks, and physical and mental health, of family caregivers of people with dementia? And, how do those health outcomes compare with similar measures for family caregivers of people with bipolar disorder? This one-year supplement study will exam these two aims as part of a larger four-year parent grant (NCT03023332). Caregivers enrolled in the study will be randomized to one of the three self-management interventions, with two data collections time points pre- and post-intervention.

DETAILED DESCRIPTION:
With every passing minute, a family member in the United States becomes an informal caregiver for an elder with Alzheimer's disease or another related dementia, which can be highly distressing and adversely affect the caregiver's mental and physical health. Similar to caregivers of persons with bipolar disorder, who are currently participating in the parent study for which this supplement is proposed, caregivers of persons with Alzheimer's or related dementia have been found to experience greater distress than caregivers of persons with other chronic conditions. They have significantly more mental and physical health problems than the general population, leading to greater use of mental health and primary care services and resulting in their inability to continue to provide care for their family members. Thus, although the trajectories of the two conditions (bipolar disorder versus dementia) may differ, we propose that caregivers of persons with dementia may benefit similarly from tailored health self-management interventions, including resourcefulness skills or biofeedback training, more than the educational materials or programs they are typically offered. Therefore, the caregivers of persons with Alzheimer's disease or related dementia to be sampled in this administrative supplement will comprise an additional study arm for the randomized controlled trial constituting the parent study. They will be randomized to: 1) usual care (education program), 2) resourcefulness training, or 3) biofeedback. Three outcomes (health risk, mental health, and physical health) will be assessed at baseline and post-intervention.

Study aims are to:

1. Examine the effectiveness of resourcefulness training and biofeedback versus usual care (education program) in family caregivers of persons with Alzheimer's disease or related dementia;
2. Compare the effects of usual care, resourcefulness training, and biofeedback obtained in caregivers of persons with dementia with those of the caregivers of persons with bipolar disorder from the parent study; and
3. Explore differences between the two types of caregivers on their needs (determined by their lowest baseline cut score on measures of knowledge, resourcefulness, and heart rate variability) and preferences (determined by asking which intervention they would have chosen) among education, resourcefulness training, or biofeedback.

Repeated measures analyses and descriptive statistics will address the study aims. Our findings will generate new scientific knowledge about the effectiveness of novel, easy to use, independently performed interventions that can be individualized and self-tailored to promote the health of Alzheimer's caregivers and other comparably distressed family caregivers.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Have a living family member with Alzheimer's disease or another dementia
* Identify self as a primary caregiver
* In-home caregivers: must be currently providing a minimum of 4 hours per day of supervision/direct care for at least the last 6 months. Caregivers whose family member lives within a facility: must report visiting their care recipient at least once per week for at least the last 6 months.
* Be capable of performing informed consent and participating in study procedures

Exclusion Criteria:

* Does not have family member with Alzheimer's disease or another dementia
* Has not cared for a living family member for at least the last 6 months.
* Has knowledge of another family member in the same household enrolled in the study
* Currently pregnant
* Has a pacemaker
* Lives outside of the study area

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2019-08-29 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaclene A Zauszniewski, PhD, Principal Investigator — Case Western Reserve University - Frances Payne Bolton School of Nursing
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 92 participants completed the informed consent process, however, 7 participants withdrew prior to the randomization process and are, consequently, excluded from the numbers below.
Period: Overall Study
Arm/Group | Biofeedback Training | Resourcefulness Training | Dementia Education
Started | 28 | 28 | 29
Received Intervention | 26 | 27 | 26
Completed | 25 | 24 | 25
Not Completed | 3 | 4 | 4
Not completed — Withdrawal by Subject | 2 | 3 | 3
Not completed — Lost to Follow-up | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All consented participants who completed T1
Groups:
- Total: Total of all reporting groups
Arm/Group | Biofeedback Training | Resourcefulness Training | Dementia Education | Total
Number analyzed (Participants) | 28 | 28 | 29 | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 15 | 15 | 44
  >=65 years | 14 | 13 | 14 | 41
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 25 | 26 | 75
  Male | 4 | 3 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 3 | 5
  Not Hispanic or Latino | 27 | 26 | 25 | 78
  Unknown or Not Reported | 1 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 7 | 7 | 23
  White | 19 | 19 | 19 | 57
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 28 | 28 | 29 | 85
Global Health [Mean (Standard Deviation); unit: units on a scale] — Measure Description: Change in Global Health - PROMIS (Patient Reported Outcomes Measurement Information System) scale. 5 items - physical health; 5 items - mental health; 5-point scale; Scores range 0-40; higher scores indicate better health.
  units on a scale | 27.21 (4.21) | 26.61 (5.26) | 27.24 (4.32) | 27.02 (4.87)
Health Risk Behavior Scale [Mean (Standard Deviation); unit: units on a scale] — Health risks were measured using the Change in Health Risk Behavior Scale. The scale consists of 9 items measured on a 3-point scale, Scores range 9-27; higher score indicates greater risk
  units on a scale | 16.12 (2.93) | 15.30 (3.27) | 14.54 (2.23) | 15.36 (2.98)
Heart Rate Variability [Mean (Standard Deviation); unit: milliseconds] — HRV is a physiological measure of the healthy functioning of the heart. It is a well-established biomarker for detecting stress. HRV was measured using the BioRadio portable limb-lead electrocardiogram recorder. Data obtained via this device was analyzed with compatible VivoSense software, which automatically computed 8 HRV parameters, including the SDNN score. The SDNN score is the standard deviation of all normal to normal R-R intervals between heartbeats and reported in milliseconds.
  milliseconds | 67.09 (57.69) | 80.22 (57.12) | 73.71 (52.95) | 73.74 (55.20)
Resourcefulness [Mean (Standard Deviation); unit: units on a scale] — Resourcefulness scale score. Composite item comprising of responses to 28 items scored on a 6 point likert scale. Scores range from 0-140, with higher scores indicating greater resourcefulness.
  units on a scale | 92.89 (15.7) | 88.29 (15.25) | 97.57 (14.72) | 92.71 (55.20)
Dementia Knowledge Scale [Mean (Standard Deviation); unit: units on a scale] — Measure of Dementia Knowledge: 25 items; true-false (5-point scale); Scores range 25-125; higher score indicates better knowledge
  units on a scale | 31.21 (8.44) | 29.18 (8.04) | 32.34 (7.40) | 30.87 (7.96)

OUTCOME MEASURES:

1. Primary Outcome: Change in Global Health - PROMIS (Patient Reported Outcomes Measurement Information System)
Description: Measure of Caregiver's Global Health: 5 items - physical health; 5 items - mental health; 5-point scale; Scores range 0-40; higher score indicates better health.
Time Frame: From T1 (baseline) through T2 (30 days post-intervention)
Population: All participants who completed both T1 and T2 questionnaires.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Biofeedback Training | Resourcefulness Training | Dementia Education
Number analyzed (Participants) | 26 | 24 | 25
score on a scale
  T1: Baseline | 27.23 (4.38) | 27.13 (4.85) | 27.52 (4.32)
  T2 | 27.23 (5.26) | 28.63 (4.56) | 28.20 (4.80)

2. Primary Outcome: Change in Health Risk Behavior Scale
Description: Measure of Caregiving Health Risks: 9 items; 3-point scale, Scores range 9-27; higher score indicates greater risk
Time Frame: From T1 (baseline) through T2 (30 days post-intervention)
Population: Includes all participants who completed both T1 and T2.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Biofeedback Training | Resourcefulness Training | Dementia Education
Number analyzed (Participants) | 26 | 24 | 25
score on a scale
  Baseline: Time 1 | 15.9 (2.80) | 14.74 (3.00) | 14.58 (2.16)
  Time 2 | 14.80 (2.82) | 15.33 (2.85) | 14.52 (2.37)

3. Secondary Outcome: Change in Dementia Knowledge Assessment Scale
Description: Measure of Dementia Knowledge: 25 items; true-false (5-point scale); Scores range 25-125; higher score indicates better knowledge
Time Frame: From T1 (baseline) through T2 (30 days post-intervention)
Population: All participants who completed both T1 and T2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Biofeedback Training | Resourcefulness Training | Dementia Education
Number analyzed (Participants) | 26 | 24 | 25
score on a scale
  Baseline: Time 1 | 31.71 (8.51) | 28.96 (7.59) | 33.52 (6.75)
  Time 2 | 33.04 (8.45) | 32.25 (6.84) | 36.28 (7.44)

4. Secondary Outcome: Change in Heart Rate Variability
Description: HRV is a physiological measure of the healthy functioning of the heart. It is a well-established biomarker for detecting stress. HRV was measured using the BioRadio portable limb-lead electrocardiogram recorder. A sensor was placed on the radial area of the caregiver's forearm for 5 minutes; they were asked to remain still as possible to prevent artifacts in the readings. The data obtained via this device was analyzed with compatible VivoSense software, which automatically computed 8 HRV parameters. One of these was the SDNN score, which is the recognized and most commonly used gold standard biomarker indicative of stress. The SDNN score is the standard deviation of all normal to normal R-R intervals between heartbeats and reported in milliseconds. The SDNN was the outcome of interest for our study as a physiological indicator of stress. For each caregiver, the software produced an average score for the 5-minute measurement
Time Frame: From T1 (baseline) through T2 (30 days post-intervention)
Population: All participants who completed both T1 and T2
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Biofeedback Training | Resourcefulness Training | Dementia Education
Number analyzed (Participants) | 26 | 23 | 25
milliseconds
  T1: Baseline | 70.60 (58.43) | 86.67 (59.14) | 79.03 (55.48)
  T2: 30 days post-intervention | 55.81 (27.22) | 43.85 (28.25) | 54.53 (33.37)

5. Secondary Outcome: Change in Resourcefulness Scale
Description: Measure of Resourcefulness: 28 items; 6-point scale; Scores range 0-140; higher score indicates more resourcefulness
Time Frame: From T1 (baseline) through T2 (30 days post-intervention)
Population: All participants who completed both T1 and T2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Biofeedback Training | Resourcefulness Training | Dementia Education
Number analyzed (Participants) | 26 | 24 | 25
score on a scale
  T1: Baseline | 91.81 (15.229) | 87.67 (16.25) | 97.20 (14.85)
  T2: 30 days post-intervention | 93.81 (15.99) | 91.08 (13.43) | 95.68 (11.79)

ADVERSE EVENTS:
Time Frame: Data was collected for the duration of the study. Participants completed a baseline questionnaire (T1), a 1 month intervention, and followup questionnaires at 6months (Q2) and 12 months (Q3) post-intervention.
Description: All events would have been reported. No adverse events occurred.
Arm/Group | Resourcefulness Training | Dementia Education | Biofeedback Training
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/29
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/47/NCT04247347/Prot_SAP_000.pdf